CLINICAL TRIAL: NCT03735745
Title: Transdisciplinary Oral/Oropharyngeal Cancer Research & Care in Head and Neck Cancer (TORCH): A Prospective Non-Randomized Study by the Head and Neck Oncology Group (HNOG) at the Medical University of South Carolina (MUSC)
Brief Title: Transdisciplinary Oral/Oropharyngeal Cancer Research & Care in Head and Neck Cancer (TORCH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 102812
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection; Tissue Banks; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Caucasian, HPV positive, Non Smoking patients (Experimental): Blood, tissue and saliva specimen will be collected. Surveys will be administered.
  Interventions: Other: Blood collection; Other: Saliva collection; Other: Tissue collection; Other: Surveys
- Caucasian, HPV positive, Smoking patients (Experimental): Blood, tissue and saliva specimen will be collected. Surveys will be administered.
  Interventions: Other: Blood collection; Other: Saliva collection; Other: Tissue collection; Other: Surveys
- Newly diagnosed, African American/Black, HPV negative, Smoking (Experimental): Blood, tissue and saliva specimen will be collected. Surveys will be administered.
  Interventions: Other: Blood collection; Other: Saliva collection; Other: Tissue collection; Other: Surveys
- Young (<40 years old), Oral Cavity (Tongue) patients (Experimental): Blood, tissue and saliva specimen will be collected. Surveys will be administered.
  Interventions: Other: Blood collection; Other: Saliva collection; Other: Tissue collection; Other: Surveys
- Neoadjuvant PD-1 Blockade patients (Experimental): Blood, tissue and saliva specimen will be collected. Surveys will be administered.
  Interventions: Other: Blood collection; Other: Saliva collection; Other: Tissue collection; Other: Surveys

INTERVENTIONS:
Other: Blood collection — 30cc of blood will be collected.
Other: Saliva collection — 5cc of saliva will be collected.
Other: Tissue collection — Up to 10mg of tissue will be collected.
Other: Surveys — The Behavioral Risk Factor Surveillance System (BRFSS), Functional Assessment of Cancer Therapy - Head and Neck module (FACT-HN) the Chicago Priority Scale, Cancer Survivor Unmet Needs surveys will be administered at baseline and 3 months post-surgery.

SUMMARY:
The purpose of this research study is to see if it is possible to collect tissue, saliva and blood samples from patients who are having surgery and send those samples to different labs across MUSC. The researchers in these labs will collect tissue, blood and saliva samples before surgery and during surgery to see if there are any changes in the samples. They will compare the changes in the samples to the clinical outcomes. Patients will also be given surveys to evaluate patient preferences, anxiety/distress, symptom severity, support by HPV status.

DETAILED DESCRIPTION:
The primary objective of this exploratory, proof of concept study is to facilitate translational science spanning clinicians and basic scientists to obtain tissue samples, PDX models, and clinical data in order to successfully analyze tissue linked to clinical outcomes in head and neck cancer, resulting in the methodological and statistical framework for a larger scale clinical trial in the future. While the incidence of HNSCC has been steadily decreasing over the last thirty years, the incidence and prevalence of oropharyngeal cancer squamous cell carcinoma (OPSCC) and young patients with oral tongue cancer has increased in the face of an overall decline in smoking prevalence. Over the past few years, evidence has emerged that oropharyngeal cancer is rising in incidence so rapidly that it has been described as an "epidemic" and that it has or soon will surpass cervical cancer in both incidence and mortality. In fact, over 30,000 patients will be diagnosed with oropharyngeal cancer in the US per year, making it the most rapidly rising head and neck cancer in incidence. Despite this unique etiopathogenesis, treatment and toxicities related to treatment have not changed. This collaboration and interdisciplinary study will be the first of its kind to address these important issues of cancer site, HPV status, tobacco history, gender, age, and race using both patient tissue and PDX models to identify novel and unique biomarkers. Also, innate to this project is the link between five separate laboratories each conducting unique biomarker analysis.

ELIGIBILITY:
Inclusion criteria:

1. Age > 18 years
2. Ability to sign informed consent
3. Newly diagnosed or recurrent oral cavity squamous cell carcinoma of the tongue (stage I-IVa) or oropharyngeal squamous cell carcinoma confirmed by pathology report. Patients with Unknown primary of the neck that is HPV+ are eligible.
4. Planning to undergo surgery as a part of definitive treatment

Exclusion criteria:

1. Squamous cell carcinoma metastasis to node(s) of neck with unknown primary tumor site that is HPV negative.
2. Already received some treatment, such as chemotherapy, radiation, or surgery for his/her disease at another institution when presenting to MUSC. An exception is neoadjuvant PD-1 blockade.
3. History of radiation therapy, for any indication, to the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Count of patients who have research blood, saliva and tissue samples collected. | 1 month (at the time of surgery)
  The number of participants to have research blood, saliva and tissues samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Besim Ogretmen, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No